CLINICAL TRIAL: NCT04855526
Title: Effects of Marijuana on Memory-Related Neurochemistry and Neural Response
Brief Title: THC + CBD and Memory Study
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Hartford Hospital (Other)
Collaborators: Yale University (Other)
Responsible Party: Principal Investigator, Godfrey Pearlson, Founding Director Olin Neuropsychiatry Research Center; Professor Yale University, Hartford Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: R-HHC-2019-0137; 126663 (Other Grant/Funding Number: Hartford Hospital)
Record Dates: First submitted 2021-04-19; First posted 2021-04-22 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Marijuana Use; Cannabis Use; Cannabis Intoxication
Keywords: marijuana; cannabidiol; memory; THC; cannabis; intoxication; MRI; glutamate; MRS
MeSH Terms: conditions — Marijuana Use; Marijuana Abuse

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Occasional Users - High THC and High CBD Dose (Experimental): People who smoke marijuana occasionally will be given a dose of high THC high CBD marijuana at the study visit
  Interventions: Drug: High THC/High CBD Marihuana
- Occasional Users - High THC and No CBD Dose (Experimental): People who smoke marijuana occasionally will be given a dose of high THC and no CBD marijuana at the study visit
  Interventions: Drug: High THC/No CBD Marihuana
- Occasional Users - No THC and No CBD Dose (Experimental): People who smoke marijuana occasionally will be given a dose of marijuana that contains no THC or CBD
  Interventions: Drug: No THC/No CBD Marihuana

INTERVENTIONS:
Drug: High THC/No CBD Marihuana — high THC (65 mg THC) and no CBD (0 mg CBD)
  Arms: Occasional Users - High THC and No CBD Dose
Drug: High THC/High CBD Marihuana — high THC (65 mg THC) and high CBD (50 mg CBD)
  Arms: Occasional Users - High THC and High CBD Dose
Drug: No THC/No CBD Marihuana — no THC (0 mg THC) and no CBD (0 mg CBD); placebo drug
  Arms: Occasional Users - No THC and No CBD Dose

SUMMARY:
Memory deficits are one of the most consistently observed cognitive effects of marijuana use. There is evidence that some decrements attributable to the primary psychoactive ingredient, delta-9-tetrahydrocannabinol (THC), may be attenuated by cannabidiol (CBD). This study will help us learn more about the relationship between THC and CBD consumption with memory processes. A combination of MRI and neuropsychological tests (which are computer and paper/pencil tasks) will be used to measure the neurocognitive and behavioral impacts of THC and CBD use.

DETAILED DESCRIPTION:
With increased legalization and medicalization of marijuana (MJ), there is an urgent need to understand the acute effects of use. One of the most consistently observed cognitive outcomes associated with MJ use is memory dysfunction, which may have a substantial impact on daily life in individuals using MJ for recreational or medicinal purposes. Notably, there are numerous preparations of MJ with varying proportions of cannabinoids, which may differ in behavioral and cognitive effects. For instance, there is emerging evidence that acute administration of delta-9-tetrahydrocannabinol (THC), the main psychoactive constituent of MJ, hinders memory and reduces prefrontal and hippocampal functional magnetic resonance imaging (fMRI) activation, but cannabidiol (CBD) may mitigate some of these impairments. Given the role of glutamate in learning and memory, the investigators suggest that these effects may be subserved, in part, by glutamatergic mechanisms. The investigators will use magnetic resonance spectroscopy (MRS) to non-invasively measure glutamate in order to explore the neurochemical underpinnings of memory-related fMRI response changes following acute administration of THC and CBD in a randomized, double-blind, placebo-controlled, cross-over design. A total of 9 healthy participants ages 18-40 will be enrolled. Participants will first undergo one screening visit (~4 hours), comprising informed consent, assessment of health history, psychiatric diagnoses, cognitive function, and substance use history, and a structural MRI session. This will be followed by 3 separate MJ dose visits (~4 hours each), at which participants will complete neuroimaging after administration of one of 3 preparations of vaporized MJ in a randomized, counterbalanced, double-blinded fashion: 1) high THC and no CBD (THC), 2) high THC and high CBD (THC+CBD), and 3) no THC and no CBD (placebo MJ). As in the investigator's ongoing studies, bulk MJ plant material will be provided by the National Institute on Drug Abuse. MJ dose visits will comprise MJ administration, blood collection, MRS/fMRI scan, subjective reports, and a brief cognitive assessment.

ELIGIBILITY:
Inclusion Criteria:

* Right-handed
* Prior MJ users (has used MJ at least once in the past year, but no more than 1x/month in the past 12 months)
* Medically healthy (as determined by medical history and treatment)
* Adequate comprehension of English in order to complete study materials
* Acceptable birth control method for women (i.e., no copper IUD or any device that is not MRI safe)

Exclusion Criteria:

* Participant currently uses psychoactive medications or substances
* Psychiatric diagnoses (determined by DSM-V)
* Participant heavily or regularly uses MJ (more than 1x/month in the past year)
* Current or past substance dependence (including MJ)
* Positive urine toxicology screens
* Positive pregnancy screens
* MRI contraindications (e.g., heart pacemaker)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
fMRI response | approximately 1 hour following drug administration
  Blood oxygen level dependent functional magnetic resonance imaging (fMRI) response during the relational and item specific encoding task. fMRI response will be evaluated during the encoding phase (relational vs. item encoding), item recognition phase (hits vs. misses for item-specific encoding, and hits vs. misses for relational encoding), and associative recognition phase (hits vs. misses).
Glutamate | approximately 1 hour following drug administration
  Magnetic resonance spectroscopy (MRS)-acquired glutamate containing compounds (Glx).

SECONDARY OUTCOMES:
HVLT-R performance | Approximately 2.50 hours after drug administration
  The Hopkins Verbal Learning Test-Revised will ascertain verbal list learning and immediate and delayed recall (~15min); alternate forms have been validated, and the order of versions participants receive will be randomized
Performance on CHARLIE cognitive task | Approximately 3.00 hours after drug administration
  This is a computer-based cognitive battery that administers the Digit Span and Letter/Number Sequencing Test (working memory) and the Digit Symbol Coding test (processing speed). It should take about 10 minutes to complete.
Blood THC and CBD concentration testing | Immediately after drug administration (~0.25 hours after drug administration)
  A blood sample will be taken once per dose visit to assess the concentration of the following metabolites in ng/mL: delta-9-tetrahydrocannabinol, 11-hydroxy-tetrahydrocannabinol, 11-Nor-9-Carboxy-tetrahydrocannabinol (THCCOOH), tetrahydrocannabinol-Glucuronide, THCCOOH-Glucuronide, cannabinol (CBN), and cannabidiol (CBD).
Subjective effects on drug effects questionnaire | Post drug administration at: 0.00 hours (immediately after); 1.0 hours; 2.0 hours; 3.0 hours
  This self-report will be used to assess subjective reports every 60 minutes throughout the dose visit days. These subjective ratings will be obtained using rapidly completed Visual Analog Scales (VASs) scored on a 0-100 scale. Items include: Do you feel a drug effect right now?, Are you high right now?, Do you dislike any of the effects you are feeling right now?, Do you like any of the effects you are feeling right now? and Would you like more of the drug you took, right now?

CONTACTS AND LOCATIONS:
Overall Officials: Godfrey Pearlson, MD, Principal Investigator — Hartford Hospital - Olin Neuropsychiatry Research Center; Yale University; Alecia Dager, PhD, Principal Investigator — Hartford Hospital - Olin Neuropsychiatry Research Center; Yale University; Michael Stevens, PhD, Principal Investigator — Hartford Hospital - Olin Neuropsychiatry Research Center

IPD SHARING:
Plan to Share IPD: No